CLINICAL TRIAL: NCT01516554
Title: A Randomized, Controlled Crossover Trial Evaluating Oral Testosterone in the Treatment of Fatigue in Male Multiple Sclerosis Patients
Brief Title: Oral Testosterone for Fatigue in Male Multiple Sclerosis Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Health Sciences Centre, Winnipeg, Manitoba (Other)
Collaborators: University of Manitoba (Other); Consortium of Multiple Sclerosis Centers (Other); Manitoba Medical Service Foundation (Other)
Responsible Party: Principal Investigator, James Marriott MD, Assistant Professor, Health Sciences Centre, Winnipeg, Manitoba
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 38486; 812.14 (Other Grant/Funding Number: Manitoba Medical Service Foundation)
Record Dates: First submitted 2012-01-19; First posted 2012-01-25 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: Multiple Sclerosis; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone undecanoate (Experimental)
  Interventions: Drug: Testosterone undecanoate
- Sugar pill (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Testosterone undecanoate — 40 mg twice daily
  Other Names: Andriol
  Arms: Testosterone undecanoate
Drug: placebo — twice daily
  Arms: Sugar pill

SUMMARY:
Fatigue is one of the most frequent symptoms reported by multiple sclerosis (MS) patients and is often a significant source of disability. Unlike normal fatigue, multiple sclerosis related fatigue (MSRF) occurs independently of activity level, suggesting that it is due to dysfunction in the neural pathways that regulate the perception of energy although the precise cause is still not understood. While MSRF can be managed through lifestyle modifications and with drug treatment, these measures are commonly either ineffective or only partially effective.

Administration of the male sex hormone testosterone has been shown to improve energy levels in males with testosterone-deficiency states. Testosterone also reduces fatigue in patients with other medical conditions not associated with low testosterone levels, suggesting that this treatment may also be useful in symptomatic control of MSRF.

This proposed seven-month long clinical trial is designed to test the hypothesis that administration of oral testosterone tablets to male MS patients will result in an improvement of fatigue relative to the administration of placebo tablets. As fatigue is frequently reported by MS patients to be one of their most frustrating and disabling symptoms, any proven additional treatment option for MSRF would be beneficial in improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All adult male (18-65 years old) patients are eligible. Patients over > 65 years will be excluded due to increased risk of prostatic hypertrophy or carcinoma in that age group.
* Patients must have diagnosis of MS using the 2005 revised McDonald Criteria.
* Patients must have an EDSS score ≤ 6.5.
* Patients must have a baseline MFIS score ≥ 45 (i.e.: those patients with fatigue).
* Patients must consent to participate in the study after a discussion of the potential risks and benefits of study participation with their physician. This consent must acknowledge that testosterone administration in MS is experimental and of no proven benefit.
* Patients must not be on any other agents to specifically treat MSRF (modafinil [Alertec®], amantadine, methylphenidate [Ritalin®, Ritalin SR®, Concerta®].

Exclusion Criteria:

* Previous or current testosterone administration.
* Any Health Canada approved indication for testosterone administration.
* Known hypersensitivity any component of the testosterone undecanoate (Andriol®) formulation including soy.
* History of relapse in the past 3 months.
* History of prostate hypertrophy or prostate carcinoma.
* History of breast cancer.
* Moderate or severe prostate symptoms (International Prostate Symptom Score [IPSS] ≥ 8).
* All patients ≥ 50 years old (or ≥ 40 years old if history of prostate cancer/prostate hypertrophy in a first-degree relative or if African-Canadian) will be require a urological assessment including prostate specific antigen (PSA) and digital rectal exam (DRE). Such patients will be excluded if they have a high PSA level or if they have a palpable prostate nodule. Abnormal PSA levels will be determined using standard age-specific cut-off levels.
* Other serious medical comorbidities including: any other cancer or myelodysplastic syndrome, anemia or polycythemia of any cause, vascular risk factors (including hypertension, dyslipidemia, myocardial infarction, stroke, peripheral vascular disease, atrial fibrillation, other hypercoaguable state or thrombotic risk factor), serious kidney or liver disease, diabetes, obstructive sleep apnea or serious psychiatric disease.
* History of current alcohol misuse.
* Recent major surgery.
* Use of the following medications whose metabolism may be altered by TT: warfarin, corticosteroids, propranolol, cyclosporine or St. John's Wort.81
* Patients on cyclophosphamide or mitoxantrone (Novantrone®) chemotherapy for MS will be excluded. Patients on other approved disease-modifying therapies for MS (interferon-β1a [Avonex®, Rebif®], interferon-β1b [Betaseron®], glatiramer acetate [Copaxone®] and natalizumab [Tysabri®]) can participate in this trial provided they have been on these therapies for at least six months at a stable dose.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in fatigue (measured with Modified Fatigue Impact Scale [M-FIS]) | baseline and 12 weeks

SECONDARY OUTCOMES:
Change in fatigue as measured on a visual analog scale (VAS) | baseline and 12 weeks
Quality of life as measured with the Aging Males' Symptoms (AMS) scale | baseline and 12 weeks
Neurological status as measured with the Expanded Disability Status Scale (EDSS) | baseline and 12 weeks
Number of participants with , type and severity of adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James J Marriott, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada